CLINICAL TRIAL: NCT02194465
Title: A Randomized, Placebo-Controlled, Double-Blinded, Parallel, Phase 2a Study to Evaluate the Safety and Efficacy of LY2623091 in Patients With Primary Hypertension
Brief Title: A Study of LY2623091 in Participants With High Blood Pressure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15525; I7T-MC-RMAH (Other: Eli Lilly and Company)
Record Dates: First submitted 2014-07-17; First posted 2014-07-18 (Estimated); Results first posted 2020-06-26 (Actual); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Primary Hypertension
MeSH Terms: conditions — Essential Hypertension | interventions — Mineralocorticoid Receptor Antagonists; Tadalafil; Spironolactone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (7):
- 6 milligrams (mg) LY2623091 (Experimental): 6 mg LY2623091 with placebo for blinding administered orally once daily for 4 weeks.
  Interventions: Drug: LY2623091; Drug: Placebo
- 13 mg LY2623091 (Experimental): 13 mg LY2623091 with placebo for blinding administered orally once daily for 4 weeks.
  Interventions: Drug: LY2623091; Drug: Placebo
- 24.5 mg LY2623091 (Experimental): 24.5 mg LY2623091 with placebo for blinding administered orally once daily for 4 weeks.
  Interventions: Drug: LY2623091; Drug: Placebo
- 13 mg LY2623091 + 20 mg tadalafil (Experimental): 13 mg LY2623091 and 20 mg of tadalafil with placebo for blinding administered orally once daily for 4 weeks.
  Interventions: Drug: LY2623091; Drug: Tadalafil; Drug: Placebo
- 20 mg tadalafil (Experimental): 20 mg tadalafil with placebo for blinding administered orally once daily for 4 weeks.
  Interventions: Drug: Tadalafil; Drug: Placebo
- Spironolactone (Active Comparator): 25 mg titrated to 50 mg as tolerated of spironolactone (open label) administered orally once daily for 4 weeks.
  Interventions: Drug: Spironolactone
- Placebo (Placebo Comparator): Placebo for blinding administered orally once daily for 4 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY2623091 — Administered orally
  Other Names: Mineralocorticoid Receptor Antagonist
  Arms: 13 mg LY2623091; 13 mg LY2623091 + 20 mg tadalafil; 24.5 mg LY2623091; 6 milligrams (mg) LY2623091
Drug: Tadalafil — Administered orally
  Other Names: LY450190
  Arms: 13 mg LY2623091 + 20 mg tadalafil; 20 mg tadalafil
Drug: Spironolactone — Administered orally
  Arms: Spironolactone
Drug: Placebo — Administered orally
  Arms: 13 mg LY2623091; 13 mg LY2623091 + 20 mg tadalafil; 20 mg tadalafil; 24.5 mg LY2623091; 6 milligrams (mg) LY2623091; Placebo

SUMMARY:
The main purpose of this study is to evaluate the safety and effectiveness of the study drug known as LY2623091 in participants with high blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Have a history of hypertension.
* If participants are naïve to treatment of hypertension, or have not been treated with any antihypertensive medications within the 30 days immediately prior to screening:

  * Have seated systolic (SBP) of ≥140 and <170 millimeters of mercury (mmHg) at screening and at the end of the lead-in period.
* If participants are currently being treated for hypertension:

  * Are taking a stable dose of 1 or 2 antihypertensive medications for at least the previous 30 days. A combination antihypertensive medication from 2 classes is considered as 2 antihypertensive medications.
  * Are willing to discontinue the antihypertensive medications during the study.
  * Have seated SBP of ≥140 and <170 mmHg at the end of the lead-in period.
* Have a body mass index (BMI) ≥18.5 and <40 kilograms/m^2.

Exclusion Criteria:

* Have a history of severe hypertension (defined as SBP ≥180 mmHg and/or diastolic (DBP) ≥120 mmHg), secondary hypertension, symptomatic postural hypotension, or hospitalization due to hypertension.
* Have SBP ≥180 mmHg and/or DBP ≥110 mmHg at screening, lead-in period, or randomization.
* Have a history of hospitalization due to hyperkalemia, or history of drug discontinuation due to elevated serum potassium levels.
* Have a serum potassium ≤3.5 or >5.0 millimoles per liter (mmol/L).
* Have an estimated glomerular filtration rate (eGFR) <50 milliliters/minute/1.73 m^2.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2014-08; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (43):
- United States (33):
  - Clinical Research Advantage, Glendale, Arizona
  - John Muir Health Network - The Osteoporosis Center, Concord, California
  - Encompass Clinical Research, Encinitas, California
  - Avail Clinical Research LLC, DeLand, Florida
  - Alan Graff, MD, PA, Fort Lauderdale, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Cardiovascular Center of Sarasota, Sarasota, Florida
  - East West Medical Institute, Honolulu, Hawaii
  - Rocky Mountain Diabetes and Osteoporosis Center, Idaho Falls, Idaho
  - Northwest Heart Clinical Research, LLC, Arlington Heights, Illinois
  - Cedar-Crosse Research Center, Chicago, Illinois
  - Midwest Institute for Clinical Research, Indianapolis, Indiana
  - Community Clinical Research Center, Muncie, Indiana
  - Heartland Research Associates, Wichita, Kansas
  - Grace Research, Bossier City, Louisiana
  - Maine Research Associates, Auburn, Maine
  - AB Clinical Trials, Las Vegas, Nevada
  - Rochester Clinical Research, Inc., Rochester, New York
  - Metrolina Internal Medicine, P.A., Charlotte, North Carolina
  - PharmQuest, Greensboro, North Carolina
  - Lillestol Research LLC, Fargo, North Dakota
  - Sterling Research Group, LTD, Cincinnati, Ohio
  - Rapid Medical Research Inc, Cleveland, Ohio
  - Columbus Clinical Research, Columbus, Ohio
  - Dayton Clinical Research, Dayton, Ohio
  - Cor Clinical Research LLC, Oklahoma City, Oklahoma
  - Oklahoma Foundation For Cardiovascular Research, Oklahoma City, Oklahoma
  - Mountain View Clinical Research, Inc, Greer, South Carolina
  - Texas Diabetes and Endocrinology, Austin, Texas
  - Tekton Research, Inc, Austin, Texas
  - Texas Diabetes and Endocrinology, P.A., Round Rock, Texas
  - Northwest Clinical Research Center, Bellevue, Washington
  - Universal Research Group, LLC, Tacoma, Washington
- Canada (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brampton
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kelowna
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Peterborough
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pointe-Claire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Québec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Red Deer
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sherbrooke
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toronto
- Puerto Rico (2):
  - Research and Cardiovascular Corp., Ponce
  - Clinical Research Puerto Rico, Inc., San Juan

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants entered at lead-in for wash out and a placebo run-in period prior to randomization.
Period: Overall Study
Arm/Group | Placebo | 6 Milligrams (mg) LY2623091 | 13 mg LY2623091 | 24.5 mg LY2623091 | 13 mg LY2623091 + 20 mg Tadalafil | 20 mg Tadalafil | Spironolactone
Started | 51 | 50 | 52 | 49 | 51 | 25 | 26
Received at Least 1 Dose of Study Drug | 51 | 50 | 51 | 49 | 51 | 25 | 26
Completed | 42 | 43 | 44 | 41 | 42 | 21 | 24
Not Completed | 9 | 7 | 8 | 8 | 9 | 4 | 2
Not completed — Adverse Event | 6 | 1 | 4 | 4 | 4 | 2 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 1 | 2 | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 3 | 1 | 2 | 2 | 1 | 2
Not completed — Discontinued follow-up period | 0 | 2 | 1 | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least 1 dose of a study drug.
Groups:
- 6 mg LY2623091: 6 mg LY2623091 with placebo for blinding administered orally once daily for 4 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | 6 mg LY2623091 | 13 mg LY2623091 | 24.5 mg LY2623091 | 13 mg LY2623091 + 20 mg Tadalafil | 20 mg Tadalafil | Spironolactone | Total
Number analyzed (Participants) | 51 | 50 | 51 | 49 | 51 | 25 | 26 | 303
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (9.4) | 56.6 (11.4) | 58.0 (8.8) | 58.7 (8.8) | 57.9 (9.5) | 54.0 (8.9) | 59.0 (11.0) | 57.7 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 17 | 24 | 20 | 21 | 8 | 7 | 113
  Male | 35 | 33 | 27 | 29 | 30 | 17 | 19 | 190
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 2 | 2 | 4 | 4 | 1 | 20
  Not Hispanic or Latino | 42 | 39 | 45 | 39 | 43 | 19 | 23 | 250
  Unknown or Not Reported | 7 | 6 | 4 | 8 | 4 | 2 | 2 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 2 | 1 | 0 | 0 | 5
  Asian | 7 | 4 | 2 | 6 | 2 | 2 | 3 | 26
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 13 | 15 | 14 | 12 | 13 | 7 | 6 | 80
  White | 28 | 30 | 34 | 29 | 35 | 15 | 16 | 187
  More than one race | 2 | 1 | 0 | 0 | 0 | 1 | 1 | 5
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 18 | 12 | 9 | 13 | 13 | 5 | 4 | 74
  United States | 32 | 36 | 41 | 35 | 38 | 19 | 21 | 222
  Puerto Rico | 1 | 2 | 1 | 1 | 0 | 1 | 1 | 7
BMI [Mean (Standard Deviation); unit: kilogram/square meter (kg/m2)] | 30.5 (4.5) | 30.2 (5.2) | 30.2 (4.9) | 32.7 (4.5) | 29.5 (4.7) | 29.6 (4.2) | 31.4 (4.5) | 30.6 (4.8)
Chronic Kidney Disease (CKD) [Count of Participants; unit: Participants]
  Y | 0 | 3 | 2 | 0 | 0 | 2 | 2 | 9
  N | 51 | 47 | 49 | 49 | 51 | 23 | 24 | 294
Anti-Hypertensive Medication [Count of Participants; unit: Participants]
  0 | 8 | 10 | 5 | 7 | 13 | 6 | 3 | 52
  1 | 24 | 22 | 25 | 22 | 17 | 10 | 10 | 130
  2 | 19 | 17 | 20 | 19 | 20 | 8 | 13 | 116
  3 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 4
  4 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Diabetes [Count of Participants; unit: Participants]
  Y | 10 | 6 | 11 | 9 | 5 | 6 | 4 | 51
  N | 41 | 44 | 40 | 40 | 46 | 19 | 22 | 252
Baseline in Seated Systolic Blood Pressure (SBP) [Mean (Standard Deviation); unit: millimeter of mercury (mmHg)] | 151.2 (8.8) | 150.8 (8.6) | 153.7 (8.3) | 150.7 (10.2) | 152.1 (9.6) | 151.7 (9.6) | 153.4 (9.0) | 151.9 (9.1)
Baseline in Seated Diastolic Blood Pressure (DBP) [Mean (Standard Deviation); unit: millimeter of mercury (mmHg)] — Population: All randomized participants receiving at least 1 dose of a study drug and had baseline seated Diastolic Blood Pressure data.
  millimeter of mercury (mmHg)
    number analyzed (Participants) | 51 | 49 | 51 | 49 | 51 | 24 | 25 | 300
    (all) | 89.8 (8.8) | 88.2 (9.7) | 90.5 (9.5) | 88.5 (8.5) | 90.6 (8.9) | 91.5 (8.8) | 88.6 (11.6) | 89.6 (9.3)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 4 Weeks in Seated Systolic Blood Pressure (SBP)
Description: Change from baseline in SBP as measured by a cuff. Least squares (LS) mean change from baseline was calculated using a mixed model repeating measures (MMRM) with treatment, country, visit, and treatment-by-visit interaction as fixed effects and baseline as a covariate.
Time Frame: Baseline, 4 Weeks
Population: All randomized participants receiving at least 1 dose of the study drug and had baseline and post baseline evaluable data for SBP.
Measure: Least Squares Mean (Standard Error); unit: millimeter of mercury (mmHg)
Arm/Group | Placebo | 6 mg LY2623091 | 13 mg LY2623091 | 24.5 mg LY2623091 | 13 mg LY2623091 + 20 mg Tadalafil | 20 mg Tadalafil | Spironolactone
Number analyzed (Participants) | 41 | 45 | 43 | 41 | 43 | 21 | 23
millimeter of mercury (mmHg) | -0.5 (11.6) | -13.1 (11.2) | -14.6 (12.3) | -14.3 (13.6) | -11.8 (12.5) | -7.1 (13.3) | -15.4 (11.7)

2. Secondary Outcome: Change From Baseline to 4 Weeks in Seated Diastolic Blood Pressure (DBP)
Description: Change from baseline in DBP as measured by a cuff. LS mean change from baseline was calculated using a MMRM with treatment, country, visit, and treatment-by-visit interaction as fixed effects and baseline as a covariate.
Time Frame: Baseline, 4 Weeks
Population: All randomized participants receiving at least 1 dose of the study drug and had baseline and post baseline evaluable data for DBP.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | 6 mg LY2623091 | 13 mg LY2623091 | 24.5 mg LY2623091 | 13 mg LY2623091 + 20 mg Tadalafil | 20 mg Tadalafil | Spironolactone
Number analyzed (Participants) | 41 | 45 | 43 | 41 | 43 | 21 | 23
mmHg | 0.5 (7.9) | -5.6 (9.2) | -4.8 (7.2) | -7.1 (7.6) | -6.8 (8.7) | -6.6 (8.7) | -1.2 (6.1)

3. Secondary Outcome: Change From Baseline to 4 Weeks in 24 Hour Ambulatory Blood Pressure Monitoring (ABPM)
Description: The LS mean change in blood pressure is calculated after adjusting for baseline, treatment and race using an analysis of covariance (ANCOVA).
Time Frame: Baseline, 4 Weeks
Population: All randomized participants receiving at least 1 dose of the study drug and had evaluable data for 24 hour ABPM.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | 6 mg LY2623091 | 13 mg LY2623091 | 24.5 mg LY2623091 | 13 mg LY2623091 + 20 mg Tadalafil | 20 mg Tadalafil | Spironolactone
Number analyzed (Participants) | 37 | 37 | 39 | 33 | 36 | 19 | 22
mmHg
  SBP | 0.3 (11.3) | -4.9 (8.7) | -11.1 (8.9) | -10.4 (11.4) | -10.4 (11.6) | -6.3 (8.9) | -6.4 (6.8)
  DBP | 1.0 (7.7) | -1.7 (6.3) | -4.7 (6.1) | -3.4 (4.8) | -6.2 (8.0) | -5.6 (4.9) | -2.0 (4.6)

4. Secondary Outcome: Change From Baseline to 4 Weeks in Serum Potassium
Description: Potassium measurement as measured by standard laboratory tests. The LS mean change in potassium is calculated using MMRM with adjustment for baseline, treatment, visit, treatment*visit and race.
Time Frame: Baseline, 4 Weeks
Population: All randomized participants receiving at least 1 dose of the study drug and had evaluable data for serum potassium.
Measure: Least Squares Mean (Standard Error); unit: millimoles/L (mmol/L)
Arm/Group | Placebo | 6 mg LY2623091 | 13 mg LY2623091 | 24.5 mg LY2623091 | 13 mg LY2623091 + 20 mg Tadalafil | 20 mg Tadalafil | Spironolactone
Number analyzed (Participants) | 42 | 45 | 43 | 41 | 44 | 21 | 24
millimoles/L (mmol/L) | -0.04 (0.06) | 0.10 (0.06) | 0.11 (0.06) | 0.25 (0.06) | 0.10 (0.06) | -0.06 (0.08) | 0.30 (0.08)

5. Secondary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY2623091
Time Frame: 2 hours post-dose at 4 Weeks
Population: All participants who had evaluable PK data of LY2623091.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter (ng/ml)
Arm/Group | 6 mg LY2623091 | 13 mg LY2623091 | 24.5 mg LY2623091 | 13 mg LY2623091 + 20 mg Tadalafil
Number analyzed (Participants) | 41 | 40 | 36 | 39
nanogram/milliliter (ng/ml) | 122 (32) | 228 (37) | 379 (51) | 206 (53)

ADVERSE EVENTS:
Description: All randomized participants who received at least 1 dose of study drug. One participant was randomized but never dosed.
Arm/Group | Placebo | 6 mg LY2623091 | 13 mg LY2623091 | 24.5 mg LY2623091 | 13 mg LY2623091 + 20 mg Tadalafil | 20 mg Tadalafil | Spironolactone
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/50 | 2/51 | 0/49 | 1/51 | 0/25 | 0/26
Other Adverse Events (participants affected / at risk) | 23/51 | 23/50 | 21/51 | 18/49 | 34/51 | 14/25 | 12/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=51) | 6 mg LY2623091 (N=50) | 13 mg LY2623091 (N=51) | 24.5 mg LY2623091 (N=49) | 13 mg LY2623091 + 20 mg Tadalafil (N=51) | 20 mg Tadalafil (N=25) | Spironolactone (N=26)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=51) | 6 mg LY2623091 (N=50) | 13 mg LY2623091 (N=51) | 24.5 mg LY2623091 (N=49) | 13 mg LY2623091 + 20 mg Tadalafil (N=51) | 20 mg Tadalafil (N=25) | Spironolactone (N=26)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bundle branch block right (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid oedema (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scleral haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Faecal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Faeces soft (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Lip swelling (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 2 (2)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Feeling abnormal (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Bronchitis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epididymitis (Infections and infestations) | 0/35 (0) | 0/33 (0) | 0/27 (0) | 0/29 (0) | 0/30 (0) | 1/17 (1) | 0/19 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 4 (4) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood potassium increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (2)
Blood pressure abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure systolic increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram t wave inversion (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heart rate increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (3) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 4 (4) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (4) | 5 (5) | 2 (2) | 1 (1) | 10 (10) | 3 (3) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tension headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0/35 (0) | 0/33 (0) | 0/27 (0) | 0/29 (0) | 1/30 (1) | 0/17 (0) | 0/19 (0)
Gynaecomastia (Reproductive system and breast disorders) | 0/35 (0) | 0/33 (0) | 0/27 (0) | 0/29 (0) | 0/30 (0) | 0/17 (0) | 1/19 (1)
Spontaneous penile erection (Reproductive system and breast disorders) | 0/35 (0) | 0/33 (0) | 0/27 (0) | 0/29 (0) | 1/30 (1) | 0/17 (0) | 0/19 (0)
Vulvovaginal dryness (Reproductive system and breast disorders) | 0/16 (0) | 1/17 (1) | 0/24 (0) | 0/20 (0) | 0/21 (0) | 0/8 (0) | 0/7 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paranasal cyst (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient acantholytic dermatosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days